CLINICAL TRIAL: NCT03109990
Title: A Pilot Study to Evaluate the Impact of Dexmedetomidine on Postoperative Tumor Recurrence in Patients With Primary Breast Cancer
Brief Title: A Pilot Study to Evaluate the Impact of Dexmedetomidine on Breast Cancer Recurrence After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DEX20161020
Record Dates: First submitted 2017-03-11; First posted 2017-04-12 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): Patients of dexmedetomidine group will receive a loading dose of 1ug/kg dexmedetomidine since 15 mins before induction, and receive another 1ug/kg of dexmedetomidine at a rate of 0.5ug/kg/h for 2 continuous hours during surgery.
  Interventions: Drug: Dexmedetomidine
- saline (Placebo Comparator): Same amount of saline will be administrated.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Patients in the experimental group will receive Dexmedetomidine during surgery.
  Arms: Dexmedetomidine
Drug: Saline — Patients in the control group will receive saline but not Dexmedetomidine during surgery.
  Arms: saline

SUMMARY:
Dexmedetomidine is widely used as an anaesthetic for general anesthesia during surgery. Previous studies in cells and animals show that dexmedetomidine may promote cancer growth. The purpose of present study is to examine whether utilization of dexmedetomidine in patients undergoing surgery for primary breast cancer increases breast cancer recurrence and metastasis, and to investigate its effects on the patients' immune system.

DETAILED DESCRIPTION:
Women diagnosed with breast cancer undergoing elective surgery under general anesthesia will be randomly allocated to dexmedetomidine group or control group. Patients from both groups will receive midazolam, propofol, fentanyl, remifentanil and CIS atracurium for total intravenous anesthesia. BIS value will be controlled between 40-60 during surgery. Patients of dexmedetomidine group will receive a loading does of 1ug/kg dexmedetomidine since 15 mins before induction, and receive another 1ug/kg of dexmedetomidine at a rate of 0.5ug/kg/h for 2 continuous hours during surgery. Patients of control group will receive same amount of normal saline. Patients will be followed up for 36 months to measure the incidence of cancer recurrence and metastasis. Serum form patients of both groups will be collected at 24 h after surgery. The number of CD3+ , CD4+, CD8+ cells and NK cells in the serum will be compared between the two groups. Serum levels of IFN-γ, IL-12，IL-4 and VEGF will also be measured and compared.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I-III
* Age range of 18 to75
* Patients diagnosed primary breast cancer
* Patients will have elective mastectomy

Exclusion Criteria:

* with history of breast operation
* Patients diagnosed with inflammatory breast
* Severe mental or physical illnesses(like liver, renal, brain or lung disease)
* with history of opioid addiction
* Patients diagnosed metastatic breast cancer
* Contradictions or an allergy to Dexmedetomidine

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
study feasibility | from May 2015 to August 2019
  recruitment and dropout rates

SECONDARY OUTCOMES:
recurrence-free survival | up to 5 years after surgery
  time from surgery to the earliest date of recurrence/metastasis
overall survival | up to 5 years after surgery
  time from surgery to the date of all-cause death
the number of blood CD3+ cells | at 24 hours after surgery
the number/percentage of blood CD4+ cells | at 24 hours after surgery
the number/percentage of blood CD8+ cells | at 24 hours after surgery
the number/percentage of blood NK cells | at 24 hours after surgery
the ratio of CD4+ cells / CD8+ cells | at 24 hours after surgery
the number/percentage of blood CD19+ cells | at 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Renji hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided